CLINICAL TRIAL: NCT01938495
Title: Multi-Center, Randomized Controlled Study of the NeuRx® Diaphragm Pacing System™ (DPS)In Participants With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Diaphragm Pacing System (DPS) In Participants With Amyotrophic Lateral Sclerosis (ALS)
Acronym: DPS in ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barrow Neurological Institute (Other)
Collaborators: ALS Association (Other); Muscular Dystrophy Association (Other); Synapse Biomedical (Industry)
Responsible Party: Principal Investigator, Jeremy Shefner, MD, PhD, Barrow Neurological Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013P001504
Record Dates: First submitted 2013-08-23; First posted 2013-09-10 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: ALS; DPS; Diaphragm Pacing
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NeuRx® Diaphragm Pacing System™ (DPS) (Experimental): Patients randomized to the experimental arm will receive The NeuRx® Diaphragm Pacing System™ (DPS) device. Under general anesthesia, the intramuscular electrodes are surgically implanted in the diaphragm.
  Interventions: Device: NeuRx® Diaphragm Pacing System™ (DPS)
- Standard of Care (No Intervention): patients randomized to the standard of care arm will not have the Diaphragm Pacing System surgically implanted but will receive standard medical care.

INTERVENTIONS:
Device: NeuRx® Diaphragm Pacing System™ (DPS) — The NeuRx® Diaphragm Pacing System™ (DPS) is a four channel, implanted percutaneous diaphragm muscle stimulation system. Pictures of the device are provided in the Clinician's Manual for the NeuRx® DPS procedure and technique guide from the manufacture Synapse Biomedical, Inc. Under general anesthesia, the intramuscular electrodes are laparoscopically implanted in the diaphragm. The ends of the implanted electrodes are tunneled subcutaneously to an exit site on the chest or abdominal wall and connected to an external stimulator.
  Arms: NeuRx® Diaphragm Pacing System™ (DPS)

SUMMARY:
The study is being conducted to determine if DPS treatment for people with ALS and hypoventilation is associated with improved survival or diaphragm function.

The primary objective of the study is to conduct a multi-center, randomized controlled clinical trial comparing standard of care (control) to diaphragm stimulator treatment with the NeuRx® Diaphragm Pacing System™ (DPS) with respect to survival.

The secondary objective of the study is to conduct a multi-center, randomized controlled clinical trial to compare standard of care treatment (control) to DPS in ALS subjects with hypoventilation.

DETAILED DESCRIPTION:
The study is a randomized controlled study to compare standard of care (control) to DPS (diaphragm stimulator named The NeuRx® Diaphragm Pacing System™). Although it remains uncertain if DPS is efficacious for the ALS subject, given the preliminary studies performed by the device manufacturer, it has received FDA humanitarian device exemption (HDE) approval as a humanitarian use device (HUD). This study will utilize a 2:1 randomization schedule such that eligible ALS subjects will have a 2/3 chance of receiving DPS and 1/3 chance of standard of care (control) treatment.

The NeuRx® Diaphragm Pacing System™ (DPS) is a four channel, implanted percutaneous diaphragm muscle stimulation system. Under general anesthesia, the intramuscular electrodes are laparoscopically implanted in the diaphragm. The ends of the implanted electrodes are tunneled subcutaneously to an exit site on the chest or abdominal wall and connected to an external stimulator.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years or older.
2. Sporadic or familial ALS diagnosed as definite, probable or possible ALS as defined by revised El Escorial criteria.
3. Evidence of hypoventilation at Screening with at least one of the following:

   1. Maximal static inspiratory pressure (MIP) <60 cm H20.
   2. Upright or supine forced vital capacity (FVC) <50% predicted for gender, age, and height.
4. A phrenic nerve potential should be recordable bilaterally.
5. Subjects must not have taken riluzole for at least 30 days, or be on a stable dose of riluzole for at least 30 days, prior to randomization (riluzole-naïve subjects are permitted in the study).
6. Capable of providing informed consent and following trial procedures.
7. Geographically accessible to the site.
8. Negative urine pregnancy test at Screening in women of child bearing potential (WOCBP). (Women who are post-menopausal or who have had a hysterectomy are deemed not of child bearing potential).
9. Women of child bearing potential must use an adequate form of contraception: abstinence, hormonal contraception (oral contraception, implanted contraception, injected contraception or other hormonal (patch or contraceptive ring, for example) contraception), intrauterine device (IUD) in place for ≥ 3 months, barrier method in conjunction with spermicide, or another adequate method.

Exclusion Criteria:

1. Upright forced vital capacity (FVC) ≤ 45% of predicted for gender, age, and height.
2. Any prior use of non-invasive ventilation (NIV) outside of sleep (nighttime or naps).
3. Any pulmonary or cardiac disorder or other medical disorder that would be a contraindication for general anesthesia or DPS hardware implantation in the chest.
4. Implanted electrical device such as a pacemaker or cardiac defibrillator.
5. Known diaphragm abnormality such as hiatal hernia or para-esophageal hernia of abdominal contents into the thoracic cavity.
6. Participation in another treatment research study for people with ALS.
7. Exposure to any other agent currently under investigation for the treatment of people with ALS (off-label use or investigational) within 30 days of the Screening Visit.
8. Clinically significant history of unstable or severe cardiac, oncologic, hepatic, psychiatric, renal disease, or other medically significant illness.
9. Pregnant women or women currently breastfeeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-08; Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Survival | Subjects will be assessed on a monthly basis for an 18 month period.

SECONDARY OUTCOMES:
quality of life | Subjects will be assessed on a monthly basis for an 18 month period.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Shefner, MD, PhD, Principal Investigator — Barrow Neurological Institute; Jonathan Katz, MD, Principal Investigator — California Pacific Medical Center
Locations (25):
- United States (25):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Diego, California
  - Stanford University, Stanford, California
  - Hospital for Special Care, New Britain, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Florida, Jacksonville, Jacksonville, Florida
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health Systems, Detroit, Michigan
  - St Louis University, St Louis, Missouri
  - Neurology Associates P.C., Lincoln, Nebraska
  - Hospital for Special Surgery, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Carolinas Health Care, Charlotte, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Providence ALS Center, Portland, Oregon
  - Drexel University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas, San Antonio, Texas
  - University of Vermont, Burlington, Vermont
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- See also: Related Info — http://alsconsortium.org